CLINICAL TRIAL: NCT04091672
Title: A Prospective Multicenter Randomized Controlled Clinical Study to Investigate the Safety and Effectiveness of the RECELL® System Combined With Meshed Autograft for Reduction of Donor Skin Harvesting in Soft Tissue Reconstruction
Brief Title: RECELL® System Combined With Meshed Autograft for Reduction of Donor Skin Harvesting in Soft Tissue Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avita Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTP007
Record Dates: First submitted 2019-09-13; First posted 2019-09-17 (Actual); Results first posted 2023-09-21 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Full-thickness Skin Defects; Degloving Injuries; Crush Injuries; Laceration of Skin; Surgical Wound; Skin Cancer; Cellulitis; Infection; Necrotizing Fasciitis; Gun Shot Wound
MeSH Terms: conditions — Degloving Injuries; Crush Injuries; Surgical Wound; Skin Neoplasms; Cellulitis; Infections; Fasciitis, Necrotizing; Wounds, Gunshot

STUDY DESIGN:
Masking Description: The participant and blinded evaluator will be not be told which treatment area received which treatment (RECELL or Control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- All Participants (within patient control) (Experimental): Each participant will serve as their own Control, receiving both Control and Investigational Interventions randomly allocated to treatment of a portion of a full-thickness skin defect.
  Interventions: Procedure: Control Intervention (Conventional Autograft); Device: Investigational Intervention (RECELL + more widely meshed autograft)

INTERVENTIONS:
Procedure: Control Intervention (Conventional Autograft) — Meshed split-thickness skin graft, with standardized wound dressings (Telfa™ Clear and Xeroform™)
  Other Names: meshed split-thickness skin graft
Device: Investigational Intervention (RECELL + more widely meshed autograft) — More widely meshed split-thickness skin graft, Spray-on Skin™ Cells prepared using RECELL, and standardized wound dressings (Telfa™ Clear and Xeroform™)

SUMMARY:
A prospective randomized within-subject controlled study to compare the clinical performance of conventional autografting with and without the RECELL system on acute non-burn full-thickness skin defects.

ELIGIBILITY:
Inclusion Criteria:

1. The patient requires autografting for treatment of an acute full-thickness skin defect (e.g., trauma- or surgery-related).
2. The maximum area requiring autografting is 50% Total Body Surface Area (TBSA).
3. Two comparable areas requiring autografting, each at least 160 cm2 (or 320 cm2 contiguous), excluding face and genitalia. When hands or joints are included in the treatment areas, comparability of treatment areas means that each area (RECELL and Control) must include the same contralateral joint and/or hand.
4. The patient is at least 5 years of age.
5. The patient (or parent/guardian) is willing and able to comply with all compulsory study procedures and visit schedule.
6. The patient agrees to abstain from any other treatment (e.g., external fixation) of the study treatment areas for the duration of his/her participation the study (1 year).
7. The patient agrees to abstain from enrollment in any other interventional clinical trial for the duration of his/her participation the study (1 year).
8. In the opinion of the investigator, the patient and/or guardian must be able to:

   1. Understand the full nature and purpose of the study, including possible risks and adverse events,
   2. Understand instructions, and
   3. Provide voluntary informed written consent.

Exclusion Criteria:

1. Not able to understand English or Spanish.
2. The area requiring autografting sustained a burn injury.
3. The treatment area has previously failed to heal subsequent to surgical intervention for closure.
4. The patient is unable to follow the protocol requirements.
5. The patient has a condition that in the investigator's opinion may compromise patient safety or trial objectives.
6. Current use of medications that in the investigator's opinion may compromise patient safety or trial objectives.
7. The patient has a known hypersensitivity to trypsin or compound sodium lactate for irrigation (Hartmann's) solution.
8. The patient is pregnant or breast-feeding (pregnancy test should be performed in accordance with local institutional requirements).
9. Life expectancy is less than 1 year.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2020-03-02 (Actual); Primary Completion 2022-03-07 (Actual); Study Completion 2023-02-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Arizona Burn Center - Valleywise Health, Phoenix, Arizona
  - University of Arizona - Banner Health, Tucson, Arizona
  - UCI Medical Center, Orange, California
  - Lundquist Institute @Harbor UCLA, Torrance, California
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Kendall Regional Medical Center, Miami, Florida
  - Cook County Health, Chicago, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - University Medical Center, New Orleans, Louisiana
  - University of Rochester Medical Center, New York, New York
  - Duke University Hospital, Durham, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Temple University, Philadelphia, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - JPS Health Network, Fort Worth, Texas
  - Metis Foundation, San Antonio, Texas

REFERENCES:
- [Derived] Henry S, Mapula S, Grevious M, Foster KN, Phelan H, Shupp J, Chan R, Harrington D, Mashruwala N, Brown DA, Mir H, Singer G, Cordova A, Rae L, Chin T, Castanon L, Bell D, Hughes W, Molnar JA. Maximizing wound coverage in full-thickness skin defects: A randomized-controlled trial of autologous skin cell suspension and widely meshed autograft versus standard autografting. J Trauma Acute Care Surg. 2024 Jan 1;96(1):85-93. doi: 10.1097/TA.0000000000004120. Epub 2023 Sep 1. PMID 38098145

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The design of this study is a within-patient comparison. Protocol enrollment is 65 (participants), with 130 interventions (2 per participant).
Units Other Than Participants: wound treatment areas
Groups:
- Control Intervention: After preparation for autografting, a portion of each participant's wound is randomly assigned to receive the Control Intervention (within-patient control).
  Conventional Autografting: Meshed split-thickness skin grafting according to a pre-specified grafting plan, along with standardized post-operative wound dressings (Telfa™ Clear and Xeroform™ wound dressings)
- Investigational Intervention (RECELL): After preparation for autografting, a portion of each participant's wound is randomly allocated to receive the Investigational Intervention.
  RECELL plus More Widely Meshed Autograft: A split-thickness skin graft meshed more widely than the pre-specified grafting plan (Control Intervention), plus RECELL, with standardized wound dressings (Telfa™ Clear and Xeroform™ wound dressings).
Period: Overall Study
Arm/Group | Control Intervention | Investigational Intervention (RECELL)
Started | 65; 65 wound treatment areas | 65; 65 wound treatment areas
Completed | 47; 47 wound treatment areas | 47; 47 wound treatment areas
Not Completed | 18; 18 wound treatment areas | 18; 18 wound treatment areas
Not completed — Death | 6 | 6
Not completed — Lost to Follow-up | 7 | 7
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Non-Compliance With Study Schedule | 2 | 2

BASELINE CHARACTERISTICS:
Population: Experimental: All Participants (within patient control)
Groups:
- Experimental: All Participants (Within Patient Control): All subjects will receive both RECELL and skin graft. Each patient serves as their own control. Their study treatment area will be divided into Area A and Area B. Investigational treatment (RECELL) will be randomly allocated to either Area A or Area B
Arm/Group | Experimental: All Participants (Within Patient Control)
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (18.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 44
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 14
  White | 46
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Treatment Area Healing
Description: The incidence of healing is hypothesized to be non-inferior for RECELL-treated areas (Investigational Intervention) as compared to Control areas (Control Intervention). Healing is defined as complete wound closure characterized by 100% skin re-epithelialization without drainage, confirmed at two consecutive study visits at least 2 weeks apart by direct visualization by a Blinded Evaluator.
Time Frame: Prior to or at 8 weeks
Population: Per protocol
Measure: Count of Units; unit: Treatment Areas
Units Other Than Participants: Treatment Areas
Arm/Group | Control Intervention | Investigational Intervention (RECELL)
Number analyzed (Participants) | 52 | 52
Number analyzed (Treatment Areas) | 52 | 52
Treatment Areas | 30 | 34
Statistical Analysis 1: Comparison: Control Intervention vs Investigational Intervention (RECELL); Test type: Non-Inferiority — The one-sided 97.5% confidence interval (97.5% CI) was calculated for the difference (Control-RECELL) in percentages of subjects with confirmed treatment area closure. The calculation used the normal approximation taking correlation into account. In order for the null hypothesis to be rejected and the non-inferiority of RECELL to be established, the upper limit of the 97.5% CI had to be less than 10%; p = .005, 1-sided z-test of proportions; alpha=0.025

2. Primary Outcome: Donor Skin Area to Treatment Area Expansion Ratio
Description: The donor skin expansion achieved with treatment using RECELL and widely meshed autograft (Investigational Intervention) is hypothesized to be superior to the donor skin expansion ratio achieved with conventional autograft treatment (Control Intervention). Expansion ratio, computed as the ratio of measured treated area to the measured donor site area, is calculated separately for each Intervention (including any donor skin needed for repeat treatments).
Time Frame: Treatment Day
Population: ITT
Measure: Mean (Standard Deviation); unit: Expansion Ratio
Units Other Than Participants: Study Areas
Arm/Group | Control Intervention | Investigational Intervention (RECELL)
Number analyzed (Participants) | 65 | 65
Number analyzed (Study Areas) | 65 | 65
Expansion Ratio | 1.39 (0.44) | 1.86 (0.47)
Statistical Analysis 1: Comparison: Control Intervention vs Investigational Intervention (RECELL); Test type: Superiority — A geometric mean ratio (GMR of ratios) 95% CI with a lower bound exceeding 1 would indicate superiority of RECELL over Control with respect to this endpoint; p = 0.001, GMR of ratios

ADVERSE EVENTS:
Time Frame: 26 Weeks
Arm/Group | Control Intervention | Investigational Intervention (RECELL)
All-Cause Mortality (participants affected / at risk) | 6/65 | 6/65
Serious Adverse Events (participants affected / at risk) | 2/65 | 2/65
Other Adverse Events (participants affected / at risk) | 35/65 | 33/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Intervention (N=65) | Investigational Intervention (RECELL) (N=65)
Impaired Healing (General disorders) | 2 (2) | 2 (2)
Local Soft Tissue Infection (Infections and infestations) | 2 (2) | 2 (2)
Other Infection (Infections and infestations) | 2 (2) | 2 (2)
Graft Loss (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin Graft Failure (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Suture Related Complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Device Malfunction (Product Issues) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Intervention (N=65) | Investigational Intervention (RECELL) (N=65)
Impaired Healing (General disorders) | 14 (14) | 12 (12)
Local Soft Tissue Infection (Infections and infestations) | 3 (4) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Graft Loss (Injury, poisoning and procedural complications) | 8 (8) | 6 (6)
Skin Graft Failure (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Skin Graft Scar Contracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Soft Tissue Foreign body (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound Decomposition (Injury, poisoning and procedural complications) | 6 (7) | 4 (4)
Wound Necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wound Secretion (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Excessive Granulation Tissue (Skin and subcutaneous tissue disorders) | 8 (8) | 12 (12)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 3 (3)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 4 (4) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT04091672/Prot_SAP_002.pdf